CLINICAL TRIAL: NCT00735540
Title: The Purpose of This Study is to Analyze the Clinical Characteristics of Teenagers Admitted to Pediatric Departments
Brief Title: Clinical Diagnosis of Teenagers Admitted to Pediatric Departments
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0022-08-EMC
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Anorexia; Thalassemia; Sickle Cell Anemia; Chronic Renal Failure; Suicide Attempt
MeSH Terms: conditions — Anorexia; Thalassemia; Anemia, Sickle Cell; Kidney Failure, Chronic; Suicide, Attempted | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- A: Acute organic diseases
  Interventions: Other: Observational
- B: Patients with chronic diseases
  Interventions: Other: Observational
- C: Patients with psychiatric diagnosis
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Data summary only

SUMMARY:
This study intends to analyze the clinical characteristics of teenagers admitted to pediatric wards due to organic illness and non organic diagnosis, including patients suffering from chronic diseases and comorbidity.

DETAILED DESCRIPTION:
The intention is to summarize the data from year 2000 to 2007 af all the teenagers aged 14 ys to 20 yes admitted to the pediatric wards at the Ha'Emek Medical Center. The demographic and clinical date will be summarized.

ELIGIBILITY:
Inclusion Criteria: All the patients ages 14 to 20 ys admitted to the pediatric ward.

Exclusion Criteria: No exclusion criteria relevant.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: About 800 teenagers are admitted each year to the pediatric departments at the Ha'Emek Medical Center. Three principal conditions are the causes of admission: chronic diseases, acute "organic" diseases, and psychiatric diseases including suicide attempts, anorexia, and others.
Sampling Method: Non-Probability Sample
Enrollment: 1389 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Analyzing the characteristics of Teenagers Admitted to Pediatric Departments | One year
  Analyzing the characteristics of Teenagers Admitted to Pediatric Departments

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit - Ha'Emek Medical Center - Afula - 18101 - Israel; Nili Gabay Saar, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center - Afula - Israel; Ziva Bracha, MD, Principal Investigator — Pediatric Psychiatric Unit - Ha'Emek Medical Center- Afula - Israel
Locations (1):
- Pediatric Dpt B - Ha'Emek Medical Center, Afula, Afula, Israel